CLINICAL TRIAL: NCT05577676
Title: Outcome Comparison of Ultrasound-guided Hydrodissection Between Normal Saline and Combination of Triamcinolone Acetonide, Normal Saline, and Lidocaine in Mild to Moderate Carpal Tunnel Syndrome: A Single Blinded Randomized Clinical Trial
Brief Title: Hydrodissection Between Normal Saline and a Combination of Triamcinolone Acetonide, Normal Saline, and Lidocaine in CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh College Of Physicians And Surgeons (BCPS) (Other)
Responsible Party: Principal Investigator, Md Mamunul Abedin, FCPS Trainee, Bangladesh College Of Physicians And Surgeons (BCPS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0161
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; CTS; Hydrodissection; Normal Saline; Triamcinolone; Ultrasound Guided
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Saline Solution; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Patients of CTS for at least 04 weeks will be selected. Informed written consent will be taken. Data will be collected by face-to-face interview. Total 62 samples will then be randomly allocated into two groups. One group will receive 5 ml of normal saline and another group will receive 5 ml combination of triamcinolone, lidocaine & normal saline. Both group will also receive Gabapentin, B vitamin, static wrist splint overnight, tendon gliding exercises and ADL advices. After taking all aseptic measures, a 23-gauze needle will be placed between transverse carpal ligament & median nerve where 3 ml fluid is given and then, at below the median nerve where another 2 ml fluid is injected. The patients will be kept in a sitting position and observed for 10 to 15 minutes before discharge.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrodissection with Normal Saline (Experimental): This group will be hydrodissected by 5 ml of normal saline, will take Gabapentin 300 mg twice daily, Neurotropic B vitamin twice daily, wear a static wrist splint in neutral position overnight, perform tendon gliding exercises 10 repetitions three times daily and maintain ADL advices.
  Interventions: Drug: Ultrasound-guided Hydrodissection of the Median Nerve
- Hydrodissection with Combination of Triamcinolone, Lidocaine, Normal Saline (Active Comparator): This group will be hydrodissected by 5 ml combination of 1 ml of triamcinolone, 1 ml of lidocaine & 3 ml of normal saline, will take Gabapentin 300 mg twice daily, Neurotropic B vitamin twice daily, wear a static wrist splint in neutral position overnight, perform tendon gliding exercises 10 repetitions three times daily and maintain ADL advices.
  Interventions: Drug: Ultrasound-guided Hydrodissection of the Median Nerve

INTERVENTIONS:
Drug: Ultrasound-guided Hydrodissection of the Median Nerve — Hydrodissection for CTS includes injecting fluid around the median nerve (MN) with 5 ml volume, 3 ml of which is given in between the transverse carpal ligament & MN, and 2 ml below the MN under Ultrasound guidance in-plane ulnar approach.
  Other Names: Ultrasound-guided Hydrodissection of the Median Nerve with Normal Saline; Ultrasound-guided Hydrodissection of the Median Nerve with Triamcinolone Acetonide

SUMMARY:
The goal of this randomized clinical trial is to compare the functional outcome of hydrodissection of the median nerve by normal saline only and a combination of triamcinolone acetonide, lidocaine, and normal saline.

The main question it aims to answer are:

• What is the outcome comparison of ultrasound-guided hydrodissection between normal saline only and combination of triamcinolone acetonide, normal saline, and lidocaine in mild to moderate carpal tunnel syndrome?

Participants diagnosed with mild or moderate CTS will be randomly assigned to two groups and be hydrodissected under ultrasound guidance.

Researchers will compare if normal saline gives similar or better functional outcomes than steroids.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is the most prevalent entrapment neuropathy caused by median nerve compression in carpal tunnel characterized by nocturnal paresthesia, tingling, numbness and pain involving glove or median distribution in hand. Almost all patients are from working group of different occupations.

The non-surgical treatments are for patients having mild to moderate CTS and these include oral steroids, drugs, braces, ultrasound therapy, tendon-gliding exercises, local steroid injection or hydrodissection etc. Hydrodissection for CTS includes injecting fluid around the nerve to eliminate the adhesions, restore blood supply and improve kinematic properties of the entrapped nerve. Ultrasound (US) - guided in-plane ulnar approach for hydrodissection in the CTS is more effective & safer. Traditionally, the steroid (triamcinolone acetonide) combined with normal saline & lidocaine is injected for this procedure. Though, the steroid injection shows greater clinical improvement only for short term, there are also possible side effects like short-lived local pain (13%), widespread axonal & myelin degeneration, skin thinning & depigmentation etc. Whereas, Normal saline (NS) is an isotonic fluid which would be suitable for expanding the perineural space. There are only a few studies comparing the outcome of hydrodissection with normal saline and triamcinolone acetonide in carpal tunnel syndrome, although the steroid injection is well established in management of CTS. Therefore, this study aims to compare the outcome between normal saline alone with combination of triamcinolone, normal saline & lidocaine. This will be a randomized clinical trial conducting in the department of Physical Medicine and Rehabilitation, Shaheed Suhrawardy Medical College Hospital, Bangladesh for 12-months period following approval of this protocol. Ethical clearance will be obtained from Ethical Review Committee (ERC) of above-mentioned hospital.

A total of 62 (sixty-two) patients above 18 years with clinical features of CTS lasting for more than 04 (four) weeks will be selected by convenience sampling and enrolled by following exclusion-inclusion criteria. All cases will be randomly assigned in to two groups (31 cases in each group) and get following treatment, i.e. Group A: Hydrodissection by 05 ml of normal saline only; Group B: Hydrodissection by 05 ml of combination of triamcinolone acetonide, normal saline & lidocaine; Both groups: Gabapentin, Neurotropic B vitamins, static wrist splint overnight, tendon gliding exercises, maintaining Activities of Daily Living (ADL) advices. Outcome will be measured by Symptom severity scale (SSS) & Functional status scale (FSS) of Boston Carpal Tunnel Questionnaire (BCQT), and Numeric pain rating score (NRS-11). Data will be taken before intervention (baseline) and 4th, 8th & 12th week after intervention. The cross-sectional area of the median nerve at carpal tunnel inlet will also be measured at the baseline & at the 12th week follow-up.

Data will be collected in a predesigned data collection sheet by face-to-face. The statistical analysis will be conducted using Statistical Package for the Social Sciences (SPSS) version 25 statistical software. The Mann-Whitney U-test and chi-square test/Fisher exact test will be used for continuous and categorical data, respectively. Intragroup data at different follow-up time-points will be evaluated using the Wilcoxon signed rank test. Differences between groups will be measured using the Mann-Whitney U-test. All statistical tests will be two-tailed, with P<0.05 considered significant. Bonferroni correction will be performed for intergroup comparisons at different time-points. All data will be presented as mean, frequency and percentages in tables, line charts etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients having pain and/or numbness, paresthesia in median nerve or glove distribution area with night symptoms for more than 4 weeks
* Patients age from 18 years of both sexes
* Electrodiagnostically (by NCS) confirmed and categorized as mild or moderate carpal tunnel syndrome
* Willing to participate

Exclusion Criteria:

* Patients having other diseases, like: Cervical radiculopathy, Other neuropathy
* History of taking systemic corticosteroids within 04-weeks prior study
* Pregnancy
* History of distal forearm or wrist fracture, trauma or deformity
* Previous CTS surgery or steroid injection in carpal tunnel
* Thenar atrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Carpal Tunnel Syndrome disease severity | 3 months
  It will be measured by Boston Carpal Tunnel Questionnaire and Numeric Pain Rating scale (NRS-11)

SECONDARY OUTCOMES:
Cross-Sectional Area (CSA) of the Median Nerve | 3 months
  It will be measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mamunul Abedin, Principal Investigator — Bangladesh College of Physicians and Surgeons
Locations (1):
- Shaheed Suhrawardy Medical College Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu PC, Liao KK, Lin KP, Chiu JW, Wu PY, Chou CL, Wang NY, Wang JC. Comparison of Corticosteroid Injection Dosages in Mild to Moderate Idiopathic Carpal Tunnel Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Nov;101(11):1857-1864. doi: 10.1016/j.apmr.2020.06.018. Epub 2020 Jul 16. PMID 32682938
- [Background] O'Connor D, Marshall S, Massy-Westropp N. Non-surgical treatment (other than steroid injection) for carpal tunnel syndrome. Cochrane Database Syst Rev. 2003;2003(1):CD003219. doi: 10.1002/14651858.CD003219. PMID 12535461
- [Background] Caliandro P, La Torre G, Aprile I, Pazzaglia C, Commodari I, Tonali P, Padua L. Distribution of paresthesias in Carpal Tunnel Syndrome reflects the degree of nerve damage at wrist. Clin Neurophysiol. 2006 Jan;117(1):228-31. doi: 10.1016/j.clinph.2005.09.001. Epub 2005 Dec 1. PMID 16325467
- [Background] Katz JN, Lew RA, Bessette L, Punnett L, Fossel AH, Mooney N, Keller RB. Prevalence and predictors of long-term work disability due to carpal tunnel syndrome. Am J Ind Med. 1998 Jun;33(6):543-50. doi: 10.1002/(sici)1097-0274(199806)33:63.0.co;2-r. PMID 9582945
- [Background] Stevens JC, Beard CM, O'Fallon WM, Kurland LT. Conditions associated with carpal tunnel syndrome. Mayo Clin Proc. 1992 Jun;67(6):541-8. doi: 10.1016/s0025-6196(12)60461-3. PMID 1434881
- [Background] Kleggetveit IP, Jorum E. Diagnosis of carpal tunnel syndrome. Scand J Pain. 2018 Jul 26;18(3):333-337. doi: 10.1515/sjpain-2018-0089. No abstract available. PMID 29894306
- [Background] Tetro AM, Evanoff BA, Hollstien SB, Gelberman RH. A new provocative test for carpal tunnel syndrome. Assessment of wrist flexion and nerve compression. J Bone Joint Surg Br. 1998 May;80(3):493-8. doi: 10.1302/0301-620x.80b3.8208. PMID 9619944
- [Background] Tai TW, Wu CY, Su FC, Chern TC, Jou IM. Ultrasonography for diagnosing carpal tunnel syndrome: a meta-analysis of diagnostic test accuracy. Ultrasound Med Biol. 2012 Jul;38(7):1121-8. doi: 10.1016/j.ultrasmedbio.2012.02.026. Epub 2012 Apr 27. PMID 22542258
- [Background] Chang KV, Wu WT, Ozcakar L. Ultrasound imaging and guidance in peripheral nerve entrapment: hydrodissection highlighted. Pain Manag. 2020 Mar;10(2):97-106. doi: 10.2217/pmt-2019-0056. Epub 2020 Mar 12. PMID 32162601
- [Background] Wu YT, Chen SR, Li TY, Ho TY, Shen YP, Tsai CK, Chen LC. Nerve hydrodissection for carpal tunnel syndrome: A prospective, randomized, double-blind, controlled trial. Muscle Nerve. 2019 Feb;59(2):174-180. doi: 10.1002/mus.26358. Epub 2018 Dec 4. PMID 30339737
- [Background] Lee JY, Park Y, Park KD, Lee JK, Lim OK. Effectiveness of ultrasound-guided carpal tunnel injection using in-plane ulnar approach: a prospective, randomized, single-blinded study. Medicine (Baltimore). 2014 Dec;93(29):e350. doi: 10.1097/MD.0000000000000350. PMID 25546691
- [Background] Kaile E, Bland JDP. Safety of corticosteroid injection for carpal tunnel syndrome. J Hand Surg Eur Vol. 2018 Mar;43(3):296-302. doi: 10.1177/1753193417734426. Epub 2017 Oct 11. PMID 29020874
- [Background] Wang PH, Tsai CL, Lee JS, Wu KC, Cheng KI, Jou IM. Effects of topical corticosteroids on the sciatic nerve: an experimental study to adduce the safety in treating carpal tunnel syndrome. J Hand Surg Eur Vol. 2011 Mar;36(3):236-43. doi: 10.1177/1753193410390760. Epub 2011 Jan 31. PMID 21282223